CLINICAL TRIAL: NCT01704547
Title: Geometric Reproducibility of the Lumpectomy Cavity Using a Breast Cup Immobilization Device II
Brief Title: Breast Cup Immobilization Device II (GCC 1047)
Acronym: BCID II
Status: Completed | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Department of Radiation Oncology, Principal Investigator, University of Maryland, Baltimore
Other Study IDs: HP-00047123
Record Dates: First submitted 2012-09-28; First posted 2012-10-11 (Estimated); Results first posted 2023-02-01 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2022-05

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Lumpectomy; Breast Irradiation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The study is designed to assess the accuracy of patient breast reproducibly using the revised BCID. This study would provide data for target verification and quality assurance to eventually allow treatment of breast cancer patients for either a TBB or accelerated partial breast irradiation. The BCID is a low-risk device similar to immobilization devices used routinely in radiotherapy for other disease sites.

DETAILED DESCRIPTION:
Breast conserving therapy (BCT) has become the standard of care for treating early-stage breast cancers based on six prospective randomized trials with 20 years of follow-up data (Fisher). During lumpectomy, the surgeon removes the tumor and a surrounding rim of normal tissue (margin), leaving surgical clips to help designate the resection bed. Radiation treatment is directed at the whole breast for 5 1/2 weeks and is generally followed by a 1-2 week boost directed at the lumpectomy site plus a margin of normal breast tissue. The benefit of adding the tumor bed boost, (TBB) has been shown in two studies to decrease local failures [Romestaig; Bartelink].

Studies have evaluated the role of radiation following lumpectomy in very select groups which have not been able to define a group who do not benefit from the addition of radiotherapy. In the group of patients who received surgery alone, 85% of the breast recurrences occurred in the tumor bed. Due to these two facts, radiotherapy directed only at the tumor bed has been evaluated. Treating this smaller tumor volume has allowed higher doses of radiation to be delivered safely shortening the treatment course from 6-7 weeks to one week.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must consent to be in the study and have signed an IRB-approved consent form.
2. The patient must have a diagnosis of invasive or non-invasive breast cancer.
3. The patient must be planned for or have already had breast conservation surgery (i.e. lumpectomy).

4 Age > 18. 5. There are at least two metal clips in the surgical cavity placed at the time of surgery for guiding the radiation oncologist in delineating the target of irradiation; or one radiographic clip placed at the time of stereotactic core needle biopsy with the intact tumor.

6. Patients who have already been treated by radiation therapy and are being seen in follow-up can also participate

Exclusion Criteria:

1. Male gender
2. Patients who cannot be set up comfortably in the prone position (e.g. physical disability)
3. Tumor/lumpectomy site located in a portion of the breast that cannot be visualized easily on the CT scan (e.g. superior portion of the upper outer quadrant).
4. Mastectomy was or is the recommended surgical approach.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer Center, Primary Care Clinic
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Nichols, MD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- Ummc Msgcc, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Breastcup: Geometric Reproducibility of the Lumpectomy Cavity Using a Breast Cup Immobilization Device II
Period: Overall Study
Arm/Group | Breastcup
Started | 25
Completed | 20
Not Completed | 5
Not completed — Physician Decision | 4
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Geometric Reproducibility of the Lumpectomy Cavity Using a Breast Cup Immobilization Device II
Arm/Group | Breastcup
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Breast Cup Immobilization Device II (GCC 1047) Feasibility
Description: Complete clinical feasibility of using a breast cup immobilization device for prone breast irradiation in terms of both geometric and dosimetric accuracy. Measurements were able to be completed on 25 participants through treatment planning CT scans.
Time Frame: One year
Population: Analysis was done through imaging assessment. Completed on all 25 patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Breastcup
Number analyzed (Participants) | 25
Participants | 25

2. Secondary Outcome: Breast Cup Immobilization Device II (GCC 1047) Comfort
Description: Assess patient comfort while wearing the breast cup immobilization device. Patients provided questionnaire to rate comfort level (discomfort was ranked from 0 (no pain) to 5 (very painful).
Time Frame: One year
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Breastcup: Assess patient comfort while wearing the breast cup immobilization device and evaluate mock treatment plans for patients using the acquired CT images.
Arm/Group | Breastcup
Number analyzed (Participants) | 25
score on a scale | 0.6 [0 to 2]

3. Secondary Outcome: Number of Participants That Were Favorable Candidates for Receiving GammaPod Treatment
Description: Candidates being assessed based on their breast size, tumor or tumor bed size, tumor or tumor bed location and normal tissue proximity by evaluating GammaPod treatment plans developed using the acquired CT images. Through images, patients were evaluated for their ability to meet the requirements for GammaPod treatment based off the factors mentioned previously.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Breastcup
Number analyzed (Participants) | 25
Participants | 25

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Breastcup
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 1/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Breastcup (N=25)
Blistering (Skin and subcutaneous tissue disorders) | 1 — Small amount (Grade 1) blistering of the skin related to suction of breast cup

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes